CLINICAL TRIAL: NCT01439022
Title: Longer-term Exercise Interventions in People With Parkinson's Disease
Brief Title: Exercise Interventions in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Royal Berkshire NHS Foundation Trust (participant identification centre) (Unknown); Nuffield Orthopaedic Centre NHS Trust (participant identification centre) (Unknown)
Responsible Party: Principal Investigator, Dr Johnny Collett, Research Fellow, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSG_EXPD_11/SC/0267
Record Dates: First submitted 2011-09-15; First posted 2011-09-22 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Exercise; Treatment Outcome; Patient Adherence
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Programme (Experimental): 6 months 2 x a week aerobic and anaerobic exercise delivered in community facilities by an exercise professional and supported by a physiotherapist.
  Interventions: Behavioral: Exercise Programme
- Hand writing programme (Active Comparator): 6 months 2 x a week hand writing practice. Performed in the home supported by a physiotherapist (5 support sessions)
  Interventions: Behavioral: Hand Writing programme

INTERVENTIONS:
Behavioral: Exercise Programme — 6 months 2 x a week aerobic and anaerobic exercise delivered in community facilities by an exercise professional and supported by a physiotherapist
  Arms: Exercise Programme
Behavioral: Hand Writing programme — 6 months 2 x a week hand writing practice. Performed in the home supported by a physiotherapist (5 support sessions)
  Arms: Hand writing programme

SUMMARY:
This study sets out to determine the effect of exercise performed over a longer period of time (6 months), delivered using community facilities, on motor and non motor symptoms, health and well being in people with Parkinson's Disease.

DETAILED DESCRIPTION:
Participation in exercise is beneficial for health and well being, but the effect over a longer period of time in people with Parkinson's disease (PD) has not been established. People with PD currently only receive short-term support for exercise therapy interventions funded from the National Health Service; it is therefore unsurprising that people with PD are observed to have low levels of physical activity that decrease over time.

Using mixed methodology the investigators will explore the effect of exercise delivered over a longer period of time (six months) in people with PD. The investigators will examine the views of people participating in the program.

Aims

Using a randomized controlled trial with one intervention arm and an active comparator control group with blinded assessments and semi-structured interview techniques the investigators will determine in people with PD:

1. The effect of longer-term exercise participation on motor symptoms
2. The effect of longer-term exercise participation on non motor symptoms, fitness, health and well being.
3. Participants views of the process and sustainability of community provision of exercise over a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosed by neurological examination; idiopathic PD defined by the UK Parkinson's Disease Society Brain Bank Criteria
* Able to walk ≥ 100m
* maintained a stable medical regime for 12 weeks prior to initiation of the study, and anticipated to maintain a stable regime for the course of study (as determined by the referring clinician).

Exclusion Criteria:

* Dementia
* History of additional prior neurological condition
* Severe depression or psychosis or a mental state that would preclude consistent active involvement with the study over its duration
* Cardiac precautions that would prevent the subject from completing the exercise program or the full battery of outcome measures
* Any known contraindication to exercise
* Reduced cognition of any cause [Minimental state examination [(MMSE) < 23]
* An orthopaedic condition that independently limits walking;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Two minute walk from baseline at 3 months | baseline and 3 months
  Distance covered in 2 minutes by walking at self selected speed
Change in Two minute walk from 3 months at 6 months | 3 months and 6 months
  Distance covered in 2 minutes by walking at self selected speed
Change in Two minute walk from 6 months at 12 months | 6 months and 12 months
  Distance covered in 2 minutes by walking at self selected speed

SECONDARY OUTCOMES:
Change in Time Up and Go (TUG) from baseline at 3 months | baseline and 3 months
  Time taken to sit to stand from a chair , walk 3 meters, turn and return to sitting in the chair. At normal speed
Change in Nine hole peg test from baseline at 3 months | baseline and 3 months
  Time taken to place 9 pegs in 9 holes and remove them
Change in SF-36 from baseline at 3 months | baseline and 3 months
  General Health status questionnaire
Change in EQ-5D from baseline at 3 months | Baseline and 3 months
  Quality of life questionnaire
Change in Prescribed medication from baseline at 3 months | baseline and 3 months
  Prescribed medication regime
Change in Blood Pressure from baseline at 3 months | baseline and 3 months
  Systolic and diastolic non-invasive blood pressure
Change in Body Mass Index from baseline at 3 months | baseline and 3 months
  Weight (kg)/ Height (m) ^2
Change in aerobic fitness from baseline at 3 months | baseline and 3 months
  An incremental cycle ergometer exercise test. (Heart rate, blood pressure, rating of perception of effort, rate of oxygen consumption (metabolism) from measures of expired air will be measured at the beginning, each increment and at the end of the test
Change in Leg power from baseline at 3 months | baseline and 3 months
  Leg power measured on the Nottingham leg power rig
Change in Grip Strength from baseline at 3 months | baseline and 3 months
  Grip strength measured by a dynamometer
Change in Disease Status from baseline at 3 months | baseline and 3 months
  Disease Status measured by Unified Parkinson's Disease Rating Scale
Change in Non-motor symptoms from baseline at 3 months | baseline and 3 months
  measured by the Non motor symptoms questionnaire
change in reported Physical Activity from baseline at 3 months | baseline and 3 months
  Self reported retrospective physical activity in social, work and home domains. Measured by the Physical Activity Scale for the Elderly questionnaire
Change measured physical activity from baseline at 3 months | baseline and 3 months
  Activity measured by an ankle worn accelerometer (steps and step intensity) over seven days
Process Evaluation | 6 months (end intervention)
  participant interviews on the perceived results and experiences/process. Interviews will be digitally audio-recorded. An interview schedule will be used to guide content. A standard thematic analysis technique will be used. The transcripts will be examined to identify themes and categories.
Adherence | Particpants will be followed at each scheduled session for the duration of the intervention (6 months 2 x a week)
  Exercise Programme: Attendance at exercise sessions and session content (Heart Rate, Rating of perceived Exertion and duration, speed and repetition of exercises)(6 months 2 x a week). Hand writing Programme: Diary of hand writing practice (6 months 2 x a week)
Change in Time Up and Go (TUG) from 3 months at 6 months | 3 months and 6 months
  Time taken to sit to stand from a chair , walk 3 meters, turn and return to sitting in the chair. At normal speed
Change in Time Up and Go (TUG) from 6 months at 12 months | 6 months and 12 months
  Time taken to sit to stand from a chair , walk 3 meters, turn and return to sitting in the chair. At normal speed
Change in Nine hole peg test from 3 months at 6 months | 3 months and 6 months
  Time taken to place 9 pegs in 9 holes and remove them
Change in Nine hole peg test from 6 months at 12 months | 6 months and 12 months
  Time taken to place 9 pegs in 9 holes and remove them
Change in SF-36 from 6 months at 12 months | 6 months and 12 months
  General Health status questionnaire
Change in SF-36 from 3 months at 6 months | 3 months and 6 months
  General Health status questionnaire
Change in EQ-5D from 3 months at 6 months | 3 months and 6 months
  Quality of life questionnaire
Change in EQ-5D from 6 months at 12 months | 6 months and 12 months
  Quality of life questionnaire
Change in Prescribed medication from 3 months at 6 months | 3 months and 6 months
  Prescribed medication regime
Change in Prescribed medication from 6 months at 12 months | 6 months and 12 months
  Prescribed medication regime
Change in Blood Pressure from 3 months at 6 months | 3 months and 6 months
  Systolic and diastolic non-invasive blood pressure
Change in Blood Pressure from 6 months at 12 months | 6 months and 12 months
  Systolic and diastolic non-invasive blood pressure
Change in Body Mass Index from 6 months at 12 months | 6 months and 12 months
  Weight (kg)/ Height (m) ^2
Change in aerobic fitness from 6 months at 12 months | 6 months and 12 months
  An incremental cycle ergometer exercise test. (Heart rate, blood pressure, rating of perception of effort, rate of oxygen consumption (metabolism) from measures of expired air will be measured at the beginning, each increment and at the end of the test
Change in Leg power from 3 months at 6 months | 3 months and 6 months
  Leg power measured on the Nottingham leg power rig
Change in Leg power from 6 months at 12 months | 6 months and 12 months
  Leg power measured on the Nottingham leg power rig
Change in Grip Strength from 3 months at 6 months | 3 months and 6 months
  Grip strength measured by a dynamometer
Change in Grip Strength from 6 months at 12 months | 6 months and 12 months
  Grip strength measured by a dynamometer
Change in Disease Status from 3 months at 6 months | 3 months and 6 months
  Disease Status measured by Unified Parkinson's Disease Rating Scale
Change in Disease Status from 6 months at 12 months | 6 months and 12 months
  Disease Status measured by Unified Parkinson's Disease Rating Scale
Change in Non-motor symptoms from 3 months at 6 months | 3 months and 6 months
  measured by the Non motor symptoms questionnaire
Change in Non-motor symptoms from 6 months at 12 months | 6 months and 12 months
  measured by the Non motor symptoms questionnaire
Change in reported Physical Activity from 3 months at 6 months | 3 months and 6 months
  Self reported retrospective physical activity in social, work and home domains. Measured by the Physical Activity Scale for the Elderly questionnaire
Change in reported Physical Activity from 6 months at 12 months | 6 months and 12 months
  Self reported retrospective physical activity in social, work and home domains. Measured by the Physical Activity Scale for the Elderly questionnaire
Change measured physical activity from 3 months at 6 months | 3 months and 6 months
  Activity measured by an ankle worn accelerometer (steps and step intensity) over seven days
Change measured physical activity from 6 months at 12 months | 6 months and 12 months
  Activity measured by an ankle worn accelerometer (steps and step intensity) over seven days
Change in FSS from baseline at 3 months | baseline and 3 months
  Fatigue measured using the FSS (Fatigue Severity Scale)
Change in FSS from 3 months at 6 months | 3 months and 6 months
  Fatigue measured using the FSS (Fatigue Severity Scale)
Change in FSS from 6 months at 12 months | 6 months and 12 months
  Fatigue measured using the FSS (Fatigue Severity Scale)
Change upper limb function from baseline at 3 months | baseline and 3 months
  upper limb function of movement time, reaction time and movement error using a touch scene PC
Change upper limb function from 3 months at 6 months | 3 months and 6 months
  upper limb function of movement time, reaction time and movement error using a touch scene PC
Change upper limb function from 6 months at 12 months | 6 months and12months
  upper limb function of movement time, reaction time and movement error using a touch scene PC

CONTACTS AND LOCATIONS:
Overall Officials: Helen Dawes, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Collett J, Franssen M, Meaney A, Wade D, Izadi H, Tims M, Winward C, Bogdanovic M, Farmer A, Dawes H. Phase II randomised controlled trial of a 6-month self-managed community exercise programme for people with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2017 Mar;88(3):204-211. doi: 10.1136/jnnp-2016-314508. Epub 2016 Nov 11. PMID 27837101
- See also: research groups website — http://www.shs.brookes.ac.uk/research/movement-science